CLINICAL TRIAL: NCT02660073
Title: Skeletal Muscle Hypertrophy and Cardio-Metabolic Benefits After Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Department of Defense (U.S. Federal Agency)
Collaborators: Hunter Holmes McGuire VA Medical Center (U.S. Federal Agency); Virginia Commonwealth University (Other); James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ashraf S. Gorgey, Director of SCI Research, Hunter Holmes McGuire VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: W81XWH-14-SCIRP-CTA
Record Dates: First submitted 2015-12-11; First posted 2016-01-21 (Estimated); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NMES+FES group (Experimental): NMES+FES group (n=24; 2 days/week for 24 weeks); this group will undergo twice weekly of 12 weeks of surface NMES and ankle weights followed by 12 additional weeks of twice weekly of progressive FES-LEC using the RT300 bike. The total participation duration is 24 weeks +3 weeks for measurements.
  Interventions: Device: NMES+FES
- Control+FES group (Experimental): Control+FES group (n=24; 2 days/week for 24 weeks); this group will undergo twice weekly of 12 weeks of passive leg extension/flexion with no ankle weights followed by 12 additional weeks of twice weekly of progressive FES-LEC using the RT300 bike. The total participation duration is 24 weeks+3 weeks for measurements.
  Interventions: Device: Control+FES

INTERVENTIONS:
Device: NMES+FES — 12 weeks of electrically evoked resistance training followed by 12 weeks of functional electrical stimulation cycling.
  Other Names: (NMES; Theratouch)+(FES; RTI300 Bike)
  Arms: NMES+FES group
Device: Control+FES — 12 weeks of passive movement followed by 12 weeks of functional electrical stimulation cycling.
  Other Names: Control+(FES; RTI300 Bike)
  Arms: Control+FES group

SUMMARY:
Spinal cord injury (SCI) is a devastating medical problem that affects thousands of civilian and military personnel in the United States. Spinal cord injuries (SCI) predispose individuals to impaired fitness, obesity, glucose intolerance and insulin resistance, placing them at greater risk for diabetes and coronary artery disease. These are devastating problems that occur frequently because of changes in body composition and reduced level of physical activity. Skeletal muscle wasting plays a central role in altered metabolism after SCI. Functional electrical stimulation (FES) is an effective rehabilitation tool that has been used to train the paralyzed skeletal muscles and which has shown some ability to ameliorate the deleterious effects of SCI on metabolism, particularly on insulin sensitivity. However, its ability to reverse skeletal muscle wasting is modest; most studies report limited gains in muscle mass and workload with highly variables outcomes from one study to another. This proposal was stimulated by the findings that a program of neuromuscular electrical stimulation resistance exercise prior to initiating functional electrical stimulation lower extremity cycling (FES-LEC) improves the gains in muscle mass and workload observed with FES. The specific objectives for the current proposal are to compare the impact of FES following evoking skeletal muscle hypertrophy of the lower extremity versus initiating FES cycling without introducing the hypertrophy effects on insulin sensitivity, control of blood sugar levels, oxygen uptake and amounts of muscle tissue and fat deposition. These studies could potentially have significant effects on thousands of people that will experience an SCI in the future as well as those living with SCI where prolonged paralysis is a major quality of life issue.

There is a major need to investigate the mechanisms lead to maximize the benefits of FES applications and to understand cellular or molecular events that are associated with muscle hypertrophy and lead to promoting metabolic health after SCI. The designed study will provide a greater understanding regarding utilization of energy sources (like fats and sugars) in muscle

DETAILED DESCRIPTION:
Primary Objectives Aim #1: To determine the impact of 12+12 weeks of neuromuscular electrical stimulation (NMES)+FES-LEC on oxygen uptake, insulin sensitivity and glucose uptake in adults with SCI compared to control + FES-LEC.

Aim #2: To determine the impact of 12+12 weeks of NMES+FES-LEC on skeletal muscle size, infiltration of intramuscular fat, visceral adiposity as well as fatigue resistance compared to control+ FES-LEC.

. Aim #3 : To determine the impact of 12+12 weeks of NMES+FES-LEC on determinants of energy metabolism, protein molecules involved in insulin signaling, muscle hypertrophy and oxygen uptake (IRS-1, adenosine monophosphate kinase (AMPK), glucose transporter (GLUT-4), insulin like growth factor (IGF-1), Akt, mammalian target of rapamycin (mTOR) and Peroxisome proliferator-activated receptor coactivator (PGC-1 alpha) and electron transport chain proteins compared to control + FES-LEC only.

Subjects: Forty eight chronic (1 year or more post-injury) individuals with motor complete SCI will be recruited from the Hunter Holmes McGuire VA Spinal Cord Dysfunction registry and Virginia Commonwealth University over 4 years.

Inclusion Criteria

1. All participants will be between 18-65 years old, men/women,
2. greater than one year post SCI,
3. Body mass index (BMI) < 30 Kg/m2.
4. Participants must have C5-L2 level of injury, traumatic motor complete or incomplete SCI [American Spinal Injury Impairment Scale Classification (AIS A, B or C)].

Exclusion Criteria:

1. Participants with any of the following pre-existing medical conditions will be excluded (cardiovascular disease, uncontrolled type II diabetes mellitus, uncontrolled hypertension, and those on insulin, pressures sores stage 3 or greater), hematocrit above 50% or urinary tract infection or symptoms.
2. Participants with osteoporosis (T-score equal or worse than -2.5 according to the World Health recommendation) will be excluded.
3. Pregnant women and women who will be involved and become pregnant during the course of the study will be excluded as well.

Study arms

1. NMES+FES group (n =24; 2 days/week for 24 weeks); this group will undergo twice weekly of 12 weeks of surface NMES and ankle weights followed by 12 additional weeks of twice weekly of progressive FES-LEC using the RT300 bike. The total participation duration is 24 weeks +3 weeks for measurements.
2. Control + FES group (n =24; 2 days/week for 24 weeks); this group will undergo twice weekly of 12 weeks of passive leg extension/flexion with no ankle weights followed by 12 additional weeks of twice weekly of progressive FES-LEC using the RT300 bike. The total participation duration is 24 weeks+3 weeks for measurements.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be between 18-65 years old,
* men/women,
* Greater than one year post SCI,
* with body mass index (BMI) < 30 Kg/m2. .
* Participants must have traumatic motor complete or incomplete SCI C5-L2 level of injury, American Spinal Injury Impairment Scale Classification (AIS A, B or C).

Exclusion Criteria:

* Participants with any of the following pre-existing medical conditions will be excluded (cardiovascular disease, uncontrolled type II DM, uncontrolled hypertension, and those on insulin, pressures sores stage 3 or greater), hematocrit above 50% or urinary tract infection or symptoms.
* Participants with osteoporosis (T-score equal or worse than -2.5 according to the World Health recommendation) will be excluded.
* Pregnant women and women who will be involved and become pregnant during the course of the study will be excluded as well.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2015-10; Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Glucose uptake | 24 weeks
  by measuring glucose effectiveness
Insulin Sensitivity | 24 weeks
  By performing frequent blood drawing of 32 samples over 3 hour period while the patient is fasting.
Oxygen Uptake | 24 weeks

SECONDARY OUTCOMES:
Skeletal Muscle Size | 24 weeks
  Magnetic Resonance Imaging
Visceral Fat | 24 weeks
  Magnetic Resonance Imaging

OTHER OUTCOMES:
Skeletal Muscle protein expressions | 24 weeks
  Muscle Biopsy of the Vastus Lateralis Muscle. The Quantity of the Protein will be determined using Western Blot.
Mitochondrial Enzyme Activities | 24 weeks
  Muscle Biopsy of the Vastus Lateralis Muscle. Mitochondrial enzyme activities will be determined using biochemical assays.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - James J. Peters VA Medical Center, The Bronx, New York
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - Virginia Commonwealth Unviersity, Richmond, Virginia

REFERENCES:
- [Derived] Gorgey AS, Venigalla S, Deitrich JN, Ballance WB, Carter W, Lavis T, Adler RA. Electrical stimulation paradigms on muscle quality and bone mineral density after spinal cord injury. Osteoporos Int. 2025 Jun;36(6):1039-1051. doi: 10.1007/s00198-025-07482-5. Epub 2025 Apr 22. PMID 40261334
- [Derived] Gorgey AS, Khalil RE, Carter W, Rivers J, Chen Q, Lesnefsky EJ. Skeletal muscle hypertrophy and enhanced mitochondrial bioenergetics following electrical stimulation exercises in spinal cord injury: a randomized clinical trial. Eur J Appl Physiol. 2025 Apr;125(4):1075-1089. doi: 10.1007/s00421-024-05661-6. Epub 2024 Nov 22. PMID 39578309
- [Derived] Gorgey AS, Khalil RE, Carter W, Ballance B, Gill R, Khan R, Goetz L, Lavis T, Sima AP, Adler RA. Effects of two different paradigms of electrical stimulation exercise on cardio-metabolic risk factors after spinal cord injury. A randomized clinical trial. Front Neurol. 2023 Sep 22;14:1254760. doi: 10.3389/fneur.2023.1254760. eCollection 2023. PMID 37808500
- [Derived] Goldsmith JA, Lai RE, Garten RS, Chen Q, Lesnefsky EJ, Perera RA, Gorgey AS. Visceral Adiposity, Inflammation, and Testosterone Predict Skeletal Muscle Mitochondrial Mass and Activity in Chronic Spinal Cord Injury. Front Physiol. 2022 Feb 10;13:809845. doi: 10.3389/fphys.2022.809845. eCollection 2022. PMID 35222077
- [Derived] Gorgey AS, Khalil RE, Davis JC, Carter W, Gill R, Rivers J, Khan R, Goetz LL, Castillo T, Lavis T, Sima AP, Lesnefsky EJ, Cardozo CC, Adler RA. Skeletal muscle hypertrophy and attenuation of cardio-metabolic risk factors (SHARC) using functional electrical stimulation-lower extremity cycling in persons with spinal cord injury: study protocol for a randomized clinical trial. Trials. 2019 Aug 23;20(1):526. doi: 10.1186/s13063-019-3560-8. PMID 31443727